CLINICAL TRIAL: NCT00028964
Title: A Randomized, Double Blind, Pacebo-Controlled Study to Assess The Feasibility, Toxicity And Efficacy (Phase I/II) Of A Chinese Herbal Therapy (CHT) For Symptom Management In Women Undergoing Chemotherapy For Stage I/II/III Breast Cancer
Brief Title: Combination Chemotherapy After Surgery With or Without Chinese Herbal Therapy to Treat Symptoms in Women With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000069154; UCSF-CRO-97755; UCSF-IND-54870; NCI-G01-2042
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer; Drug/Agent Toxicity by Tissue/Organ
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; recurrent breast cancer; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Cyclophosphamide; Doxorubicin; Chemotherapy, Adjuvant

INTERVENTIONS:
Dietary Supplement: Chinese herbs
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Herbs used in traditional Chinese medicine may decrease the side effects of chemotherapy.

PURPOSE: Randomized phase I/II trial to study the effectiveness of herbs used in traditional Chinese medicine in decreasing the side effects of chemotherapy after surgery in women who have stage I, stage II, or early stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects and safety of chinese herbal therapy (CHT) when administered for toxicity attenuation in combination with adjuvant doxorubicin and cyclophosphamide in women with stage I, II, or early stage III breast cancer.
* Determine patient compliance and the feasibility of using CHT by daily treatment calendars, weekly symptom inventories, and quality of life and mood state questionnaires completed by these patients.
* Determine patient preferences and concerns about CHT.
* Determine, preliminarily, the efficacy of CHT in ameliorating the toxic effects/side effects of adjuvant chemotherapy with doxorubicin and cyclophosphamide, in terms of the incidence and severity of adverse events, in these patients.

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive adjuvant doxorubicin IV and cyclophosphamide IV over 1 hour on days 0, 21, 42, and 63. Patients also receive oral chinese herbal therapy three times daily on days -10 to 105.
* Arm II: Patients receive adjuvant chemotherapy as in arm I and oral placebo three times daily on days -10 to 105.

Quality of life is assessed at baseline and on days 3, 24, 45, 66, 84, and 105.

Patients are followed at day 105.

PROJECTED ACCRUAL: A total of 60 patients (30 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I, II, or early stage III breast cancer for which adjuvant doxorubicin and cyclophosphamide is recommended
* No metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Over 18

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 9.0 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 2 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No evidence of acute ischemic cardiac disease on ECG

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of multiple severe food or medicine allergies or sensitivities
* No medical or psychological condition that would preclude study participation
* No severe concurrent illness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 3 weeks since prior investigational agents
* At least 3 weeks since prior herbal therapy
* No other concurrent investigational agents
* No other concurrent herbal therapy or alternative medicine
* Concurrent acupuncture allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States